CLINICAL TRIAL: NCT04750200
Title: Management of Chronic Subdural Hematoma With or Without Embolization of Middle Meningeal Artery in Canada (EMMA-Can)- A Randomized Control Trial.
Brief Title: Management of CSDH With or Without EMMA- a Randomized Control Trial
Acronym: EMMA-Can
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Jai Shankar, Professor, Department of Radiology, Neuro-Interventional Radiologist, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS24435 (B2020:120)
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Subdural Hematoma
Keywords: chronic subdural hematoma, Embolization of Middle Meningeal artery (EMMA)
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Intervention Model Description: open-label randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Patients randomized to the control arm will undergo institutional standard of care treatment (surgical drainage) for the CSDH.
- Interventional Arm (Experimental): Patients randomized to the interventional arm will undergo institutional standard of care treatment (surgical drainage) for the CSDH followed by EMMA within 72 hours of surgical drainage. The embolization will be done using a liquid embolic agent (Onyx) and will be done under a general anesthesia or conscious sedation as per the operator's preference. All patients will be followed as per the institutional standard of the care. Any peri-procedural complications and change in clinical status will be recorded.
  Interventions: Procedure: Embolization of the Middle Meningeal Artery

INTERVENTIONS:
Procedure: Embolization of the Middle Meningeal Artery — EMMA is performed inside of the blood vessels where tiny catheters are used to deliver a liquid embolic agent (Onyx) to block small blood vessels supplying the brain coverings.
  Arms: Interventional Arm

SUMMARY:
EMMA-Can is a prospective randomized open-label, blinded end point (PROBE) study, that will assess the recurrence risk and safety of embolization of the middle meningeal (EMMA) when added to standard of care treatment (surgical drainage) of chronic subdural hematoma (CSDH) compared to surgical treatment alone.

DETAILED DESCRIPTION:
All patients in clinical need of surgical drainage for the CSDH will be randomized in our study. Patients that present in the Emergency Department (ED) or neurosurgery clinic will be assessed for standard of care treatment options based on their presenting symptoms. Patients will then by screened for study eligibility based on the study inclusion and exclusion criteria. After screening and consenting patients will be randomized in to the control arm or interventional arm.

Patients randomized to the control arm will receive institutional standard of care treatment (surgical drainage) of the CSDH.

Patients randomized to the interventional arm will receive institutional standard of care treatment (surgical drainage) of the CSDH followed by EMMA, with Onyx and under a general anesthetic within 72 hours of surgical drainage.

All patients will be followed as per the institutional standard of the care. Any peri-procedural complications and change in clinical status will be recorded. The risk of recurrence at 90-days will be assessed in all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Premorbid Modified Rankin Scale of ≤2;
2. Patients with unilateral symptomatic primary or recurrent CSDH >10 mm in thickness on CT head undergoing surgical drainage;
3. CT Angiogram of head and neck which favors vascular access for EMMA and lacks dangerous anatomic variations;
4. Patients over 18 years of age; no upper age limit.

Exclusion Criteria:

1. If informed consent cannot be obtained from the patients or their substitute decision makers;
2. Patients with bilateral symptomatic CSDH;
3. CTA showing persistent communication between branches of middle meningeal artery and that of internal carotid arteries;
4. Contraindication to the embolization procedure such as severe renal dysfunction (eGFR<30), or pregnancy;
5. Life expectancy < 6 months;
6. Known allergy to Onyx;
7. Acute subdural hematoma with homogenous hyperdensity on CT scan;
8. Secondary CSDH that may likely be due to the underlying condition such as a vascular lesion, brain tumor, arachnoid cyst, spontaneous intracranial hypotension or prior craniotomy;
9. Patients needing treatment with 2 weeks of dexamethasone or tranexamic acid will be contraindicated in the study patients to avoid confounding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Subdural Hematoma (CSDH) recurrence at 90-days on CT scan | 90-days
  Symptomatic recurrence of the CSDH on CT scan of head within 90-days from EMMA

SECONDARY OUTCOMES:
90 day mRs ≤3 | 90-days
  Percentage of patients with a Modified Rankin score ≤3.
Reduction of CSDH size at 90-days | 90-days
  Reduction of the size of the CSDH on CT scan of the head at 90 days from EMMA.
Mortality within 90-days | "up to 90-days"
  Peri-procedural mortality related to EMMA
Morbidity within 90-days | " up to 90-days"
  Peri-procedural morbidity related to EMMA such as, puncture site hematoma, arterial dissection or stroke
90-day MOCA and EQ-5D-5L health score | " Day 90"
  Score on the Montreal Cognitive Assessment test and score on the EQ-5D-5L assessment
Discharge destination | "Discharge Day"
  Discharge location from acute care
Length of hospital stay | "Discharge Day"
  Number of days of acute care hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jai JS Shankar, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No